CLINICAL TRIAL: NCT06571266
Title: A Phase 1 Pharmacokinetic Study in Healthy Subjects to Evaluate the Relative Bioavailability of Two Formulations of Risankizumab Following Subcutaneous Administration With Prefilled Syringes
Brief Title: A Study to Assess the Relative Bioavailability of Two Formulations of Risankizumab Following Subcutaneous Administration With Prefilled Syringes in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M24-342
Record Dates: First submitted 2024-08-23; First posted 2024-08-26 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; Risankizumab; ABBV-066
MeSH Terms: interventions — risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Risankizumab Formulation 1 (Experimental): Participants will receive a single dose of Risankizumab formulation 1 on day 1.
  Interventions: Drug: Risankizumab
- Risankizumab Formulation 2 (Experimental): Participants will receive a single dose of Risankizumab formulation 2 on day 1.
  Interventions: Drug: Risankizumab
- Risankizumab Formulation 3 (Experimental): Participants will receive a single dose of Risankizumab formulation 3 on day 1.
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Risankizumab — • Subcutaneous Injection via prefilled syringe
  Other Names: ABBV-066; SKYRIZI

SUMMARY:
This study will assess the pharmacokinetics, relative bioavailability and tolerability of two formulations of risankizumab following subcutaneous (SC) administration in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Body weight 40 kg to 100 kg, inclusive, at screening and upon initial confinement
* Body Mass Index (BMI) is > = 18.0 to < = 32.0 kg/m2 after rounded to the tenths decimal, at Screening and upon confinement.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead ECG.

Exclusion Criteria:

* Participant with exposure to any anti-interleukin-12/23 or anti-interleukin-23 treatment for at least one year prior to Screening.
* Participant with intention to perform strenuous exercise within at least one week prior to administration of study drug or during the study.
* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 231 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to day 140
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Maximum Observed Serum Concentration (Cmax) of Risankizumab | Up to Day 140
  Cmax will be assessed of Risankizumab
Time to Cmax (Tmax) of Risankizumab | Up to Day 140
  Tmax will be assessed of Risankizumab
Apparent Terminal Phase Elimination Rate Constant (β) of Risankizumab | Up to Day 140
  Apparent terminal phase elimination rate constant (β) will be assessed of Risankizumab
Terminal Phase Elimination Half-life (t1/2) of Risankizumab | Up to Day 140
  Terminal phase elimination half-life (t1/2) will be assessed of Risankizumab
Area Under the Concentration-time Curve (AUC) from Time 0 to Time of the Last Measurable Concentration (AUC0-t) | Up to Day 140
  AUC0-t will be assessed
AUC from Time 0 to Infinity (AUC0-inf) of Risankizumab | Up to Day 140
  AUC0-inf will be assessed of Risankizumab
Number of Anti-drug antibody (ADA) Titers | Up to Day 140
  Incidence and concentration of anti-drug antibodies

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (3):
- United States (3):
  - Cenexel Act /ID# 270310, Anaheim, California
  - Collaborative Neuroscience Research CNS /ID# 270286, Los Alamitos, California
  - Acpru /Id# 270152, Grayslake, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-342